CLINICAL TRIAL: NCT06504108
Title: Evaluation Of The Efficacy Of Using Calcium-Silicate Based Sealers As A Pulp Capping Material After Adult Pulpotomy: An In-vivo Study
Brief Title: Full Pulpotomy Procedure of Permanent Molar Teeth of Adults Using Calcium Silicate-based Sealer Material
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mahmoud Yahia Ramadan Abdelsalam, Master Degree in Endodontics, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 959/1498
Record Dates: First submitted 2024-06-18; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Irreversible Pulpitis
Keywords: pulpotomy; calcium silicate-based sealer; irreversible pulpitis; MTA

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- calcium silicate-based sealer (Experimental): Performing full pulpotomy of permanent mandibular and maxillary molar teeth using calcium silicate-based sealer as a capping agent.
  Interventions: Procedure: Calcium silicate-based sealer full Pulpotomy
- Premixed calcium silicate-based putty (Active Comparator): Performing full pulpotomy of permanent mandibular and maxillary molar teeth using premixed calcium silicate-based putty as a capping agent.
  Interventions: Procedure: Calcium silicate-based premixed putty full Pulpotomy
- combination between calcium silicate-based sealer and premixed calcium silicate-based putty (Experimental): Performing full pulpotomy of permanent mandibular and maxillary molar teeth using a combination of calcium silicate-based sealer and premixed calcium silicate-based putty as a capping agent.
  Interventions: Procedure: Full Pulpotomy

INTERVENTIONS:
Procedure: Calcium silicate-based sealer full Pulpotomy — Using calcium silicate-based sealer as a capping agent after full pulpotomy
  Arms: calcium silicate-based sealer
Procedure: Calcium silicate-based premixed putty full Pulpotomy — Using calcium silicate-based premixed putty as a capping agent after full pulpotomy
  Arms: Premixed calcium silicate-based putty
Procedure: Full Pulpotomy — Using combination between calcium silicate-based sealer and calcium silicate-based premixed putty as a capping agent after full pulpotomy
  Arms: combination between calcium silicate-based sealer and premixed calcium silicate-based putty

SUMMARY:
This clinical study aims to assess the efficacy of using calcium silicate based sealer as a capping material after complete removal of coronal pulp tissue. The study will evaluate both the clinical and radiographic changes.

DETAILED DESCRIPTION:
Root canal treatment has always been considered the first line of treatment for carious teeth with symptomatic irreversible pulpitis for a long time. However, after the evolution of calcium silicate based materials a more conservative option, which is pulpotomy began to gain reliability, especially that it preserves the vitality of the radicular pulp, clinically simpler, less time-consuming, and more cost-effective compared to conventional root canal treatment.

In this study the investigators assess the clinical and radiographic success rate of using calcium silicate based sealer as a pulp capping material in permanent molars after pulpotomy.

For the best of the investigators' knowledge, there is no available clinical data on the use of calcium-silicate based sealers as a pulp capping material in pulpotomy of permanent molars with symptoms of irreversible pulpitis.

ELIGIBILITY:
Inclusion Criteria:

* Vital mandibular molar teeth with mature apices.
* Teeth that respond positively to cold testing.
* Teeth without any signs of necrosis including sinus tract or swelling.
* Teeth with caries extending ≥ 2/3 of dentine or exposing the pulp.
* Teeth with symptomatic irreversible pulpitis with/without apical periodontitis.
* Teeth without periodontal diseases or mobility.
* Teeth without root resorption, detectable pulp chamber and root canal calcification or history of trauma.
* Patients from both genders with age range from 20 to 45 years old.
* Patients with good or moderate oral hygiene and without any systemic diseases.

Exclusion Criteria:

Pre-operative criteria:

* Non-vital teeth.
* Teeth with irreversible pulpitis with apical periodontitis.
* Teeth with immature apices.
* Teeth with Periodontal disease or mobility grade II or III.
* Teeth that are badly decayed and need post and core placement.
* Patients refused to continue treatment procedures or refuse to commit to periodic follow-up sessions.
* Non-restorable teeth.

Intra-operative criteria:

* If hemostasis could not be achieved within 6 minutes after full pulpotomy.
* Teeth with partial necrosis.
* No bleeding after access cavity preparation.

Post-operative criteria:

* presence of Swelling.
* presence of Sinus tract.
* Pain on percussion after the end of the first week.
* Pain with palpation.
* Pain on biting after the end of first week.
* Mobility of the tooth.
* Fracture of tooth structure that renders the tooth non-restorable.
* Fracture of the restoration during the evaluation.
* Probing depth more than 3 mm.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Clinical success after full pulpotomy procedure | immediate postoperative
  Clinical evaluation of the targeted tooth is performed and the treatment is considered successful in case of: absence of post-operative pain, absence of pain on percussion and palpation, absence of any swelling related to the treated tooth, absence of sinus tract or fistula and absence of tooth mobility.
Radiographic success after full pulpotomy procedure | immediate postoperative
  Radiographic evaluation of the targeted tooth is performed and the treatment is considered successful in case of presence of normal periodontal ligament space, absence of internal or external root resorption, absence of canal calcification, absence of peri-radicular radiolucency and no loss or break of lamina dura.
Clinical success after full pulpotomy procedure | At 1 month
  Clinical evaluation of the targeted tooth is performed and the treatment is considered successful in case of absence of post-operative pain, absence of pain on percussion and palpation, absence of any swelling, absence of sinus tract or fistula and absence of tooth mobility.
Cinical success after full pulpotomy procedure | At 3 months
  Clinical evaluation of the targeted tooth is performed and the treatment is considered successful in case of: absence of post-operative pain, absence of pain on percussion and palpation, absence of any swelling related to the treated tooth, absence of sinus tract or fistula and absence of tooth mobility.
Clinical success after full pulpotomy procedure | At 6 months
  Clinical evaluation of the targeted tooth is performed and the treatment is considered successful in case of: absence of post-operative pain, absence of pain on percussion and palpation, absence of any swelling related to the treated tooth, absence of sinus tract or fistula and absence of tooth mobility.
Radiographic success after full pulpotomy procedure | At 6 months
  Radiographic evaluation of the targeted tooth is performed and the treatment is considered successful in case of presence of normal periodontal ligament space, absence of internal or external root resorption, absence of canal calcification, absence of peri-radicular radiolucency and no loss or break of lamina dura.
Clinical success after full pulpotomy procedure | At 9 months
  Clinical evaluation of the targeted tooth is performed and the treatment is considered successful in case of: absence of post-operative pain, absence of pain on percussion and palpation, absence of any swelling related to the treated tooth, absence of sinus tract or fistula and absence of tooth mobility.
Clinical success after full pulpotomy procedure | At 12 months
  Clinical evaluation of the targeted tooth is performed and the treatment is considered successful in case of: absence of post-operative pain, absence of pain on percussion and palpation, absence of any swelling related to the treated tooth, absence of sinus tract or fistula and absence of tooth mobility.
Radiographic success after full pulpotomy procedure | At 12 months
  Radiographic evaluation of the targeted tooth is performed and the treatment is considered successful in case of presence of normal periodontal ligament space, absence of internal or external root resorption, absence of canal calcification, absence of peri-radicular radiolucency and no loss or break of lamina dura.

SECONDARY OUTCOMES:
Assessment of Post-operative pain after full pulpotomy procedure | 6 hours, 24 hours, 48 hours, 72 hours and 7 days
  The postoperative pain was assessed by using the modified verbal descriptor Scale (mVDS). Patients were instructed to place a mark on the horizontal scale to represent the intensity of pain experienced, furthermore, they were asked to use the verbal descriptors as a guide. The level of pain was documented at the range of 0-10 numerically and verbally as no pain (0), slight pain (1, 2), moderate pain (3-5), strong pain (6, 7), severe pain (8), and maximum pain (9, 10).

CONTACTS AND LOCATIONS:
Overall Officials: Moataz A Elkhawas, PhD, Study Chair — Faculty of Dental Medicine, Al-Azhar University, Cairo
Locations (1):
- Faculty of Dental Medicine, Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
I am planning to share the study protocol and clinical study report
Supporting Information: Study Protocol, CSR
Time Frame: Once I get the Results
Access Criteria: Full access to the selected data

REFERENCES:
- [Background] Taha NA, Al-Khatib H. 4-Year Follow-up of Full Pulpotomy in Symptomatic Mature Permanent Teeth with Carious Pulp Exposure Using a Stainproof Calcium Silicate-based Material. J Endod. 2022 Jan;48(1):87-95. doi: 10.1016/j.joen.2021.09.008. Epub 2021 Sep 24. PMID 34563506
- [Background] Asgary S, Eghbal MJ, Shahravan A, Saberi E, Baghban AA, Parhizkar A. Outcomes of root canal therapy or full pulpotomy using two endodontic biomaterials in mature permanent teeth: a randomized controlled trial. Clin Oral Investig. 2022 Mar;26(3):3287-3297. doi: 10.1007/s00784-021-04310-y. Epub 2021 Dec 2. PMID 34854987
- [Background] Asgary S, Eghbal MJ, Fazlyab M, Baghban AA, Ghoddusi J. Five-year results of vital pulp therapy in permanent molars with irreversible pulpitis: a non-inferiority multicenter randomized clinical trial. Clin Oral Investig. 2015 Mar;19(2):335-41. doi: 10.1007/s00784-014-1244-z. Epub 2014 Apr 27. PMID 24771228
- [Background] Eghbal MJ, Asgary S, Baglue RA, Parirokh M, Ghoddusi J. MTA pulpotomy of human permanent molars with irreversible pulpitis. Aust Endod J. 2009 Apr;35(1):4-8. doi: 10.1111/j.1747-4477.2009.00166.x. PMID 19335509
- [Background] Lin LM, Ricucci D, Saoud TM, Sigurdsson A, Kahler B. Vital pulp therapy of mature permanent teeth with irreversible pulpitis from the perspective of pulp biology. Aust Endod J. 2020 Apr;46(1):154-166. doi: 10.1111/aej.12392. Epub 2019 Dec 21. PMID 31865629
- [Background] Tzanetakis GN, Koletsi D, Georgopoulou M. Treatment outcome of partial pulpotomy using two different calcium silicate materials in mature permanent teeth with symptoms of irreversible pulpitis: A randomized clinical trial. Int Endod J. 2023 Oct;56(10):1178-1196. doi: 10.1111/iej.13955. Epub 2023 Jul 26. PMID 37452640
- [Background] Taha NA, Abuzaid AM, Khader YS. A Randomized Controlled Clinical Trial of Pulpotomy versus Root Canal Therapy in Mature Teeth with Irreversible Pulpitis: Outcome, Quality of Life, and Patients' Satisfaction. J Endod. 2023 Jun;49(6):624-631.e2. doi: 10.1016/j.joen.2023.04.001. Epub 2023 Apr 19. PMID 37080387